CLINICAL TRIAL: NCT07056790
Title: Research on the Application of 68Ga-PSMA-CYC PET Imaging in the Diagnosis, Staging, and Restaging of Prostate Cancer
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Fujian Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAHFJ-68Ga-PSMAcyc
Record Dates: First submitted 2025-06-30; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Prostate CA
Keywords: psma; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients will undergo a 68Ga-PSMA-CYC PET/CT 、68Ga-PSMA-617 or 68Ga-PSMA-11 PET/CT (Active Comparator): Prostate Patients received 68Ga-PSMA-CYC 、68Ga-PSMA-617 or 68Ga-PSMA-11 PET/CT imaging within one week. Tracer doses of 68Ga-PSMA-CYC、68Ga-PSMA-617 or 68Ga-PSMA-11 will be used to image lesions of prostate cancer by PET/CT
  Interventions: Drug: 68Ga-PSMA-CYC
- 68Ga-PSMA-CYC (Experimental): Experimental: dynamic PET scans PET imaging will begin at 3 minutes, 15 minutes, 30min minutes, 60 minutes and 150 minutes after injection
  Interventions: Drug: CYC

INTERVENTIONS:
Drug: 68Ga-PSMA-CYC — Each prostate cancer patient underwent a 68Ga-PSMA-CYC (3-4 mCi) PET/CT scan, as well as a 68Ga-PSMA-617 (3-4 mCi) or 68Ga-PSMA-11 (3-4 mCi) PET/CT scan, with the time interval between the two scans not exceeding one week.
  Arms: Patients will undergo a 68Ga-PSMA-CYC PET/CT 、68Ga-PSMA-617 or 68Ga-PSMA-11 PET/CT
Drug: CYC — The dose will be 3-4mCi given intravenously.
  Arms: 68Ga-PSMA-CYC

SUMMARY:
68Ga-PSMA-CYC is a novel radiotracer targeting PSMA. In this study, we investigated the safety, biodistribution, radiation dosimetry of 68Ga-PSMA-CYC PET/CT in patients with prostate cancer, and performed a head-to-head comparison with 68Ga-PSMA-617 and 68Ga-PSMA-11 to evaluate its diagnostic performance.

DETAILED DESCRIPTION:
Prostate cancer (PCa) is one of the most common malignant tumors among men worldwide. Prostate-specific membrane antigen (PSMA) is a transmembrane glycoprotein that is highly expressed in PCa and its metastatic lesions, making it an ideal target for the precise diagnosis and treatment of PCa. Various low-molecular-weight radiopharmaceuticals targeting PSMA have been developed, such as PSMA-11 and PSMA-617, which can be labeled with 68Ga or 177Lu. 68Ga-PSMA-CYC is a novel radiotracer that has demonstrated favorable in vivo and in vitro stability in preliminary studies, with specific accumulation in PCa, high binding affinity, and good safety profile, making it a promising candidate for further investigation. This prospective study aims to investigate the safety, biodistribution, radiation dosimetry of 68Ga-PSMA-CYC PET/CT in patients with prostate cancer, and performed a head-to-head comparison with 68Ga-PSMA-617 and 68Ga-PSMA-11 to evaluate its diagnostic performance.

ELIGIBILITY:
Inclusion Criteria:

* confirmed treated or untreated prostate cancer patients;
* signed written consent.

Exclusion Criteria:

* known allergy against PSMA;
* any medical condition that in the opinion of the investigator may significantly interfere with study compliance.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Diagnostic value | through study completion, an average of 1year
  Sensitivity and Specificity of 68Ga-PSMA-CYC for prostate cancer in comparison with 68Ga-PSMA-617 and 68Ga-PSMA-11 PET/CT.
Adverse events | Within 7 days following PET/CT
  The safety will be assessed by the number and percentage of patients with adverse events; Adverse events were categorized using the Common Toxicity Criteria for Adverse Events 5.0.

SECONDARY OUTCOMES:
Dosimetry data | through study completion, an average of 3 months
  Calculate the absorbed dose of 68Ga-PSMAcyc in normal organs.

CONTACTS AND LOCATIONS:
Overall Officials: Weibing Miao, MD, Principal Investigator — First Affiliated Hospital of Fujian Medical University
Locations (1):
- The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No